CLINICAL TRIAL: NCT04057053
Title: Netarsudil Use After Descemetorhexis Without Endothelial Keratoplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Emma C. Davies, MD, Assistant Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-101H; 2019P000908 (Other: MGB IRB)
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Fuchs' Endothelial Dystrophy; Cataract
Keywords: DWEK, Netarsudil
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract | interventions — netarsudil; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a pilot study to determine whether there is any benefit to using Netarsudil after DWEK surgery. The study plans to enroll 10 patients (20 eyes) with Fuchs endothelial dystrophy and cataract to under combined cataract surgery with DWEK sequentially in both eyes. The first eye will be treated with Netarsudil after surgery and time to clearance will be noted. The second eye will not be treated with Netarsudil and if time to clearance is longer than the first eye, Netarsudil will be added to test if it can be used as a "rescue" drop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Netarsudil use (Experimental): Patient eye undergoes cataract surgery + DWEK, immediately after surgery Netarsudil 0.02% ophthalmic 1 drop daily is used in the operative eye until corneal clearance is documented.
  Interventions: Drug: Netarsudil 0.02% Ophthalmic Solution
- Standard of care + possible rescue drop (Active Comparator): Patient eye undergoes cataract surgery + DWEK, no Netarsudil is used after surgery, if cornea is not cleared in time for first eye Netarsudil 0.02% ophthalmic 1 drop dailyadded daily as possible rescue drop and time to corneal clearance is documented
  Interventions: Drug: Netarsudil 0.02% Ophthalmic Solution

INTERVENTIONS:
Drug: Netarsudil 0.02% Ophthalmic Solution — Use of Netarsudil 0.02% ophthalmic solution daily after surgery

SUMMARY:
Primary aim of the study is to determine whether a rho kinase inhibitor, Netarsudil, can speed corneal clearance after DWEK. Secondary aim of the study is to investigate whether patient factors, such as baseline age, pachymetry, or endothelial cell count influence response to Netarsudil.

DETAILED DESCRIPTION:
Spontaneous corneal clearance after Descemetorhexis without keratoplasty (DWEK) has been documented in several previous trials. One of the largest cohorts at Massachusetts Eye and Ear Infirmary demonstrated spontaneous corneal clearance in about 82% of cases but mean time to clearance was approximately three months after the procedure. During this time period, patients have significantly reduced central vision. Furthermore, some patients fail to have corneal clearance even eight months after DWEK and have to undergo Descemet membrane endothelial keratoplasty (DMEK) to achieve corneal clearance. A recent international case report has documents that the addition of a rho kinase inhibitor, Ripasudil, to two eyes that failed to clear by two to three months after DWEK resulted in corneal clearance within two weeks after the addition of Ripasudil. This finding indicates the possibility that a rho kinase inhibitor can be used to speed corneal clearance after purposeful Descemetorhexis. The only FDA approved rho kinase inhibitor eye drop currently available is Netarsudil, approved in December of 2017 for use in ocular hypertension and primary open angle glaucoma. Investigating whether Netarsudil can speed corneal clearance after DWEK is truly importance as the potential to expand patient eligibility for DWEK is significant. Both patients that had previously not wanted to wait approximately three months after the procedure for corneal clearance as well as patients with lower mid-peripheral endothelial cell counts may now be eligible for a procedure to treat corneal endothelial dysfunction without a corneal transplant. This would reduce risks for corneal transplant rejection and failure, reduce need for long-term steroid eye drop use, and reduce need for frequent corneal screenings to ensure transplant health.

The current study aims to investigate whether the off-label use of Netarsudil can improve corneal clearance after DWEK in Fuchs endothelial dystrophy patients.

ELIGIBILITY:
Inclusion Criteria:

* Cataract in both eyes
* Fuchs endothelial dystrophy in both eyes

Exclusion Criteria:

* History of ocular surgery in one eye and not the other
* History of significant ocular trauma/burn in one eye and not the other
* Inability to provide informed consent
* Inability to undergo eye surgery
* Inablity to use eye drops reliably

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Time to corneal clearance | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emma E Davies, Principal Investigator — Massachusetts Eye and Ear Infirmary; Roberto Pineda, Principal Investigator — Massachusetts Eye and Ear Infirmary; Ula Jurkunas, Principal Investigator — Massachusetss Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No